CLINICAL TRIAL: NCT06567405
Title: Impact of Derma Pen in the Treatment of Gingivitis Induced by Orthodontic Therapy
Brief Title: Derma Pen as Treatment of Gingivitis Induced by Orthodontics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Safa Basiouny Alawy (Other)
Responsible Party: Sponsor-Investigator, Safa Basiouny Alawy, Lecturer of Orthodontics, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #R-OMPDR-5-24-3111
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gingivitis; Orthodontic Appliance Complication
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I: dermapen and topical ascorbic Acid (Experimental): 12 individuals who have orthodontically induced gingivitis will be treated with dermapen and topical ascorbic Acid
  Interventions: Device: Derma pen with topical ascorbic Acid
- group II: mechanical periodontal treatment (Active Comparator): 12 individuals who have orthodontically induced gingivitis will receive mechanical periodontal treatment only
  Interventions: Procedure: mechanical periodontal treatment

INTERVENTIONS:
Procedure: mechanical periodontal treatment — Patients will undergo subgingival scaling employing a Piezoelectric ultrasonic scaler to eliminate local factors.
  Arms: group II: mechanical periodontal treatment
Device: Derma pen with topical ascorbic Acid — local anesthesia of 2% lignocaine will be administered by infiltration technique in the anterior maxillary region. Microneedling of the mucosa will be performed using dermapen needles, employing an intermittent back-and-forth motion in the anterior maxillary and mandibular region for 30-40 seconds, reaching a depth of 1.5 mm. This will involve the creation of microholes in the gingival tissue using derma pen to enhance the concentration and penetration of the ascorbic Acid through the gingival tissues.
  Arms: group I: dermapen and topical ascorbic Acid

SUMMARY:
Although orthodontic therapy frequently improves tooth alignment and appearance, its problems with oral hygiene can make patients highly susceptible to gingivitis. After orthodontic treatment, gingivitis is a typical problem. New treatments that promote healing and decrease inflammation are needed. Ascorbic acid and Derma Pen used together have recently surfaced as a potentially effective therapy option for patients who seeking for periodontal therapy during and after orthodontic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. patients age: 18-25 years .
2. systemically healthy patients.
3. mild to moderate plaque-induced gingivitis patients during orthodontic therapy

Exclusion Criteria:

1. periodontitis.
2. individuals who smoke or those who have tobacco related habits.
3. partially edentulous individuals.
4. individuals who are diagnosed with drug-induced gingival enlargement.
5. Pregnant or lactating women

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
gingival index (GI) | one month
  gingival index will be calibrated using William's probe approximately 1 to 2 mm to the margin of the gingiva at an angulation of 45 degree to document the gingival inflammation signs of the upper six anterior teeth. Each of the four surfaces of the anterior teeth (buccal, lingual, mesial, and distal) will be given a score from 0 to 3 and then areas were added and divided by four to give the accurate GI of each tooth.
  Score 0 = No signs of inflammation, bleeding, or swelling. Score 1= Presence of signs of mild inflammation, slight edema, and color change but no bleeding.
  Score 2 = Presence of moderate inflammation, redness, swelling, and bleeding on probing.
  Score 3 = Presence of severe inflammation, marked redness, edema, and spontaneous bleeding.

SECONDARY OUTCOMES:
Plaque Index (PI) | one month
  PI will be measured to record soft deposit accumulations on the upper six anterior teeth. Each of the four surfaces of the anterior teeth (buccal, lingual, mesial, and distal) will be given a score from 0 to 3 and then areas were added and divided by four to give the accurate PI of each tooth.
  Sore 0 = No plaque. Score 1 = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after using the probe on the tooth surface (not seen by the naked eye).
  Score 2 = Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eye.
  Score 3 = Abundance of soft deposits within the gingival pocket and/or on the tooth and gingival margin that covers the interdental areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Tanta, Egypt